CLINICAL TRIAL: NCT03854864
Title: Evaluation by Oncologists of Strategies for the Prevention and Treatment of Chemotherapy-induced Peripheral Neuropathies: Observational and Cross-sectional Study
Brief Title: Evaluation by Oncologists of Strategies for the Prevention and Treatment of Chemotherapy-induced Peripheral Neuropathies
Acronym: EVANEURO
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UFR de Pharmacie (Clermont-Ferrand) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-426
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Peripheral Nervous System Diseases; Oncologists
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncologists: French oncologists
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — to assess the current practices of management by oncologists in France in 2019, for any type of practitioners of university hospital, or general hospital, for all type of neurotoxic anticancer drugs.

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is one of the most deleterious adverse effect of neurotoxic anticancer drugs affecting up to 40% of patients. These neurotoxic anticancer agents include mainly: cisplatin (bronchopulmonary cancers), oxaliplatin (colorectal cancers), paclitaxel (breast cancers and bronchopulmonary cancers), docetaxel (breast cancers and bronchopulmonary cancers) and bortezomib (multiple myeloma).

CIPN affects not only the quality of life of patients, it also has a major impact on oncology strategy, forcing oncologists to reduce dose-intensity, to stop an ongoing chemotherapy regimen and to change therapeutic strategies, with a risk of compromising patients' survival.

There is no real preventive or curative treatment (except duloxetine) for CIPN and it is not known what is the practice of oncologists in France? However, it is essential to know the degree of sensitivity of oncologists to this problem and their practice.

With this study, the investigators propose to assess the current practices of management by oncologists in France in 2019, for any type of practitioners of university hospital, or general hospital, for all type of neurotoxic anticancer drugs.

DETAILED DESCRIPTION:
This observational and cross-sectional study will be conducted as a survey using the REDCap software and the response to this survey will be done online, in real time, with an automatic, secure and centralized data collection (CHU Clermont-Ferrand).

French oncologist will be contacted by email thanks to the regional cancer networks. Answer to the survey will be done online.

ELIGIBILITY:
Inclusion Criteria:

* Oncologist

Exclusion Criteria:

* pain physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: oncologist
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Treatment strategy for CIPN | at day 1
  Name of the drug used to treat CIPN and therapeutic adjustments, relay to a pain doctor and use of drugs)

SECONDARY OUTCOMES:
Perception of effectiveness of the treatments used | at day 1
  Visual analogic scale: 0 no efficacy - 100 maximal efficacy
Perception of safety of the treatments used to treat CIPN | at day 1
  Visual analogic scale: 0 unacceptable adverse effect - 100 acceptable adverse effects
Treatment strategy for CIPN prevention | at day 1
  Name of the drug used to prevent CIPN and therapeutic adjustments
Estimation by the oncologist of the percentage of patients affected by CIPN | at day 1
  Visual analogic scale: 0% - 100% of patients
Proportion of assessments of the CIPN severity performed by the oncologist using a specific questionnaire | at day 1
  yes / no (percentage) if yes name of the questionnaire
Proportion of CIPN assessments performed by the oncologist with a clinical examination | at day 1
  yes / no (percentage)
Proportion of CIPN assessments performed by a neurological examination (neurologist) | at day 1
  yes / no (percentage)
Age of oncologists | at day 1
  years
Sex of oncologists | at day 1
  Male / female
Organ or system speciality of oncologists | at day 1
  name of speciality
Number of chemotherapy prescriptions | at day 1
  Number of chemotherapy
Types of neurotoxic anticancer drugs prescribed | at day 1
  Name of drugs
Working place | at day 1
  French region of practice and type of structure (public / private)

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Selvy M, Pereira B, Kerckhove N, Busserolles J, Farsi F, Guastella V, Merle P, Pezet D, Balayssac D. Prevention, diagnosis and management of chemotherapy-induced peripheral neuropathy: a cross-sectional study of French oncologists' professional practices. Support Care Cancer. 2021 Jul;29(7):4033-4043. doi: 10.1007/s00520-020-05928-6. Epub 2021 Jan 5. PMID 33403401